CLINICAL TRIAL: NCT02972944
Title: Acute Cholecystitis in the Elderly: Comparative Randomized and Cohort Study of Laparoscopic Cholecystectomy vs. Conservative Treatment With Antibiotics Alone
Brief Title: Laparoscopic Cholecystectomy or Conservative Treatment in the Acute Cholecystitis of Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Tampere University Hospital (Other); Oulu University Hospital (Other); Mikkeli Central Hospital (Other); North Karelia Central Hospital (Other); Jyväskylä Central Hospital (Other); Päijänne Tavastia Central Hospital (Other); Central Hospital of Hämeenlinna (Unknown); Central Hospital of Jorvi (Unknown)
Responsible Party: Principal Investigator, Hannu Paajanen, Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 326/2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-25 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-02

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecystectomy group (Experimental): Cholecystectomy group will undergo laparoscopic cholecystectomy within 48 hrs after randomization.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Non-operative group (Active Comparator): Patients of non-operative group will be treated conservatively with intravenous antibiotics (cefuroxime) at surgical ward. Elective cholecystectomy will not be arranged.
  Interventions: Procedure: Non-operative treatment

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy
  Arms: Cholecystectomy group
Procedure: Non-operative treatment
  Arms: Non-operative group

SUMMARY:
Cholecystectomy is the only curative treatment for gallstone disease of acute calculous cholecystitis.The purpose of this study is to find the most effective treatment (laparoscopic cholecystectomy vs. conservative) for elderly patients with acute cholecystitis. Therefore a randomized multi-centre study of 200 elderly patients suffering from acute cholecystitis is performed with additional cohort of all elderly patients with acute cholecystitis in the study hospitals during study period.

DETAILED DESCRIPTION:
The increasing age is one of the main risk factors for developing complicated gallstone disease. Currently, there is lack of good quality studies comparing risks and benefits of early laparoscopic cholecystectomy in the elderly patients. Cholecystectomy is the only curative treatment for gallstone disease of acute calculous cholecystitis.

Aim: The purpose is to find out the most effective treatment (laparoscopic cholecystectomy vs. conservative) with the least morbidity for elderly patients with acute cholecystitis.

Study design: multicenter randomized controlled trial (RCT) and additional cohort of all elderly patients (>75 years old) with acute cholecystitis.

Patient allocation: Elderly patients with diagnosis of acute cholecystitis will be randomly allocated to either early laparoscopic cholecystectomy or treatment with antibiotics. Reasonably healthy elderly patients (ASA 2-3) are included in this study, excluding the patients with ASA-class above 4.

Interventions: The study group of patients will undergo early laparoscopic cholecystectomy within 48 hours after hospitalization. The control group will be managed conservatively with intravenous antibiotics and elective cholecystectomy will not be scheduled later.

Primary outcome: Assessment of morbidities related to acute cholecystitis and individual quality of life. Secondary outcomes include number of hospital admissions, length of hospitalization, pain, complications, mortality and cost analysis.

Sample size and data-analysis: Based on data of previous studies the recruitment of 200 patients in total is expected. Follow-up will be for 12 months.

In addition of RCT, we decided to record and analyze all acute cholecystitis of elderly patients in study hospitals during the study period. We will present these results in the connection of RCT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed acute cholecystitis
* Age over 75 yrs
* American Association of Anesthesiologists Classification class 2-3
* Duration of symptoms < 5 days

Exclusion Criteria:

* American Association of Anesthesiologists Classification class 4-5
* Age under 75 yrs
* Peritonitis
* Sepsis or septic shock
* Duration of symptoms over 6 days
* Cholestasis or diagnosed stone at common biliary duct.
* Acute Pancreatitis

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Specific Morbidity Index Scores | 1 year postoperatively
  The primary outcome is morbidity, all complications will be scored (according to "morbidity-index" -chart) (ref: Gutt et al: Ann Surg 2013;258:385-393)

SECONDARY OUTCOMES:
Quality of life RAND-36 scores | pre-operatively and 1 year postoperatively
  Quality of life according to RAND-36
Pain scores (0-100) | pre-operatively, 1 week, 1 month and 1 year postoperatively
  Pain (VAS, range 0-100)
Number of patients with failure of antibiotic therapy | 1 week, 1 month and 1 year postoperatively
  Recurrent cholecystitis after antibiotic therapy
Time of hospitalization (days) | 1 month
  Length of time at hospital
Mortality (number of patients) | 1 month
  Death within 30 d
Number of patients with complications | 1 week, 1 month and 1 year postoperatively
  Bile duct injury, re-operations, bile leakage, hemorragia, wound infections, pneumonia etc.
Cost analysis in euros | 1 week, 1 month and 1 year postoperatively
  cost analysis comparison between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No